CLINICAL TRIAL: NCT03383393
Title: Pharmacologic Treatment of Myocardial Ischemia Detected by Intracoronary ECG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexandrovska University Hospital (Other)
Responsible Party: Principal Investigator, Lyubomir Dosev, Doctor, Principal Investigator, Alexandrovska University Hospital
Other Study IDs: Alexandrovska UH
Record Dates: First submitted 2017-12-04; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Coronary Ischemia
MeSH Terms: interventions — Eptifibatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- adenosine: Intracoronary bolus of adenosine (adenocor)
  Interventions: Drug: Intracoronary bolus of adenosine (adenocor), Integrilin (eptifibatide) or nitroglyzerin (nitronal)
- GP IIb/IIIa: Intracoronary bolus of Integrilin (eptifibatide)
  Interventions: Drug: Intracoronary bolus of adenosine (adenocor), Integrilin (eptifibatide) or nitroglyzerin (nitronal)
- Nitroglycerine: Intracoronary bolus of nitroglycerine (nitronal)
  Interventions: Drug: Intracoronary bolus of adenosine (adenocor), Integrilin (eptifibatide) or nitroglyzerin (nitronal)

INTERVENTIONS:
Drug: Intracoronary bolus of adenosine (adenocor), Integrilin (eptifibatide) or nitroglyzerin (nitronal) — intracoronary drugs

SUMMARY:
After PCI searching for target lesion ischemia with intracoronary ECG will be performed and if found it will be treated pharmacologically

DETAILED DESCRIPTION:
The study will include patients with coronary lesions and PCI. It will include patients with stable or unstable angina, without elevated hs-TnT. PCI will be performed and monitoring of intracoronary ST elevation. Any dissection or acute vessel closure will be promptly treated with balloon or stenting.

Although there could be good angiographic result sometimes ischemia could be detected in the treated region by means of intracoronary ECG ST elevation above 1mm.

This study aims to tackle this issue with randomization of the patients into three possible treatments - intracoronary adenosine, IIb/IIIa inhibitors or nitroglycerine alone - intracoronary ST segment will be searched for reverse or residual ischemia after the pharmacologic bolus.

The intracoronary electrocardiography (i.c. ECG) is a very sensitive method for ischemia detection. The i.c. ECG reacts earlier on ischemia; the changes are much more prominent and easy to register. The wire tip could be positioned directly in different regions and thus to "map" regional ischemia. In most of the studies and from our own observations became evident that when surface ECG do not react the i.c. ECG demonstrates significant changes in ST-segment and QRS complex. Moreover, the registration of i.c. ECG is very cheap and needs only an adapter connecting coronary wire end and ECG. An i.c. ECG also can differentiate residual ischemic changes in distal main vessel and side branch as sources of prolonged ischemia, respectively - source of periprocedural myonecrosis.

Once good angiographic result is obtained after stenting there could be different reasons for ischemia in the treated region - microembolic debris or coronary microvascular spasm.

ELIGIBILITY:
Inclusion Criteria:

* Subject at least 18 years of age.
* Target lesion(s) located in a native coronary artery with diameter of ≥ 2.5 mm and ≤ 4.5 mm. If there is side branch lesion(s) located in a native coronary artery with diameter of ≥ 2.0 mm.
* Target lesion(s) amenable for PCI with balloon angioplasty of the side branch.

Exclusion Criteria:

* Subjects with significant ST-T change (≥ 1mm).
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Subjects who refuse to give informed consent.
* Subjects with the following angiographic characteristics: left main coronary artery stenosis, total occlusion target lesion, lesion of interest located at infarct-related artery.
* Subjects with LVEF < 30%.
* Subjects with moderate or severe degree valvular heart disease or primary cardiomyopathy.
* LBBB, RBBB, atrial fibrillation/flutter with no identifiable isoelectric line.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that go under percutaneous interventions
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01-03 (Estimated); Primary Completion 2019-12-05 (Estimated); Study Completion 2019-12-05 (Estimated)

PRIMARY OUTCOMES:
Intracoronary ischemia change after intracoronary drug bolus | 12 months
  Look for ischemia change after intracoronary drugs

SECONDARY OUTCOMES:
Target lesion revascularization | 12 months
  Any revascularization at the territory of previously implanted stent.
Number of patients not alive | 12 months
  death
Myocardial infarction | 12 months
  MI after discharge
New onset angina or heart failure symptoms | 12 months
  New onset angina symptoms of at least CCS class II; New onset dyspnea at exertion or at rest

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandrovska University Hospital, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided